CLINICAL TRIAL: NCT03464734
Title: An Open Label, Single-arm, Phase 2 Study of Pembrolizumab and Nanoparticle Albumin-bound Paclitaxel in Patients With Metastatic Urothelial Carcinoma After Chemotherapy Failure; the PEANUT Study
Brief Title: Pembrolizumab and Nab Paclitaxel in Patients With Metastatic Urothelial Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEANUT
Record Dates: First submitted 2018-02-19; First posted 2018-03-14 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Metastatic Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — pembrolizumab; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab + nab-paclitaxel (Experimental): pembrolizumab 200 mg + nab-paclitaxel 125 mg/m2, intravenously
  Interventions: Drug: Pembrolizumab and Nanoparticle Albumin-bound Paclitaxel

INTERVENTIONS:
Drug: Pembrolizumab and Nanoparticle Albumin-bound Paclitaxel — At study entry, patients will receive 2 cycles of pembrolizumab at the dose of 200 mg, intravenously in 30 min, on day 1 and nab-paclitaxel 125 mg/m2 intravenously in 30-40 min, on day 1 and 8.

SUMMARY:
This phase II, single-center study will assess the efficacy of pembrolizumab + nab-paclitaxel in patients who have metastatic urothelial tumor and do not respond to chemotherapy. The time between drug administration and progression of the disease will be assessed to determine if the drug will work.

DETAILED DESCRIPTION:
In an open-label, single-arm, single-center, phase 2 trial, patients will receive pembrolizumab 200 mg intravenously (IV) on D1 and nab paclitaxel at the dose of 125 mg/m2 IV on D1 and D8. Cycles are repeated every 3 weeks until PD or onset of unacceptable toxicity. Key inclusion criteria are: predominant UC, failure of maximum 2 platinum-based CT regimens for metastatic disease (2nd-to-3rd line only). Neoadjuvant/adjuvant CT is counted if relapse occurred 6 months of the last CT cycle. Response is evaluated by RECIST criteria v.1.1 every 2 cycles. PD-L1 expression will be prospectively assessed on both immune cells (IC) and tumor cells at a centralized laboratory (National Cancer Institute Milano). Combined positivity score (CPS) for PD-L1 assessment will be used, as previously reported, and the 10% cutoff will be adopted for the analyses. The primary endpoint of the study is the progression-free survival (PFS). The target is to detect an improvement in the median PFS from 3.0 months (H0) to 5.0 months (H1). To achieve 90% power with a one-sided non-parametric test at the 10% significance level, we estimated that 64 patients must be accrued over 18 months, with follow-up duration of 12 months. PFS will be also analyzed according to the PD-L1 expression. Should the above investigation suggest that the treatment benefit is stronger in patients with CPS 10%, there is the option to expand this cohort up to a maximum of 50 patients. As such, we estimate 85% power to detect the target improvement in PFS. The decision of cohort expansion will rely on predictive power (PP) calculation: a PP 30% will be regarded as promising. Translational analyses will include multiparametric flow cytometry of blood samples, gene expression (RNA-seq, Illumina HiSeq) and mutation profiling of tumor samples (Ion Torrent Personal Genome Machine). These profiles will be matched with response to treatment and PFS/overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial, and be willing and able to follow trial procedures.
2. Be 18 years-old on day of signing informed consent.
3. Have an histologically-confirmed diagnosis of UC of the bladder or the urothelium, originating from either the bladder or the urinary tract (including upper tract), with predominant (>50%) UC component if other divergent histologies (e.g. squamous cell carcinoma, adenocarcinoma, small cell carcinoma) are found.
4. Have a life expectancy of at least 12 weeks.
5. Have experienced failure of 1 or 2 platinum-based conventional chemotherapy regimens for metastatic disease (2nd-to-3rd line only); a relapse should be occurred within 6 months from the last cycle of chemotherapy.
6. Have measurable disease based on RECIST 1.1.
7. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may provide an archived specimen.
8. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
9. Demonstrate adequate organ function.
10. (Female subject of childbearing potential) Have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
11. (Female subjects of childbearing potential ) Be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication.
12. (Male subjects of childbearing potential) Agree to use an adequate method of contraception, starting from the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
3. Has a known history of active Bacillus Tuberculosis
4. Had prior administration of taxane-based chemotherapy
5. Is taking regular oral steroids, above the allowed limit of 10mg/day methylprednisolone or analogues, for any reason. Patients must not have had steroids for 28 days prior to study entry
6. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., Grade ≤1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
7. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent

   * Note: Subjects with Grade ≤2 neuropathy are an exception to this criterion and may qualify for the study
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
8. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
9. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
11. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
12. Has an active infection requiring systemic therapy.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
16. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
17. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies)
18. Has known active Hepatitis B or Hepatitis C
19. Has received a live vaccine within 30 days of planned start of study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2020-01-21 (Actual)

PRIMARY OUTCOMES:
Progression-free-survival | Through study completion, average 4 months
  Increment of median PFS from 3 months to 5 months, with 10% of statistical significance

SECONDARY OUTCOMES:
Incidence of all-grade and grade 3-4 side effects | 9 weeks
  number of patients with adverse events, frequency and type of adverse events
Objective response-rate (ORR) to RECIST v1.1 criteria | 9 weeks
  Rate of complete response + partial response
Overall survival | Through study completion, average 6 months
  overall survival

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Clinical Trial Center, Istituto Nazionale dei Tumori di Milano, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Giannatempo P, Raggi D, Marandino L, Bandini M, Fare E, Calareso G, Colecchia M, Gallina A, Ross JS, Alessi A, Briganti A, Montorsi F, Madison R, Necchi A. Pembrolizumab and nab-paclitaxel as salvage therapy for platinum-treated, locally advanced or metastatic urothelial carcinoma: interim results of the open-label, single-arm, phase II PEANUT study. Ann Oncol. 2020 Dec;31(12):1764-1772. doi: 10.1016/j.annonc.2020.09.012. Epub 2020 Sep 23. PMID 32979512
- See also: Pembrolizumab and nab-paclitaxel as salvage therapy for platinum-treated, locally advanced or metastatic urothelial carcinoma: interim results of the open-label, single-arm, phase II PEANUT study — https://pubmed.ncbi.nlm.nih.gov/32979512/